CLINICAL TRIAL: NCT06583993
Title: A Clinical Trial Assessing the Safety and Efficacy of Intravenous HNF4α srRNA for the Treatment of Patients With Advanced Intrahepatic Cholangiocarcinoma
Brief Title: A Clinical Trial Evaluating the Safety and Efficacy of Intravenous HNF4α srRNA in Treating Advanced ICC Patients
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai Changzheng Hospital (Other)
Responsible Party: Principal Investigator, Wei-Fen Xie, Director, Department of Gastroenterology, Changzheng Hospital, Shanghai Changzheng Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CZXH-ICC-2024-IIT-2
Record Dates: First submitted 2024-08-28; First posted 2024-09-04 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Intrahepatic Cholangiocarcinoma
Keywords: Intrahepatic Cholangiocarcinoma; Hepatocyte nuclear factor 4α
MeSH Terms: conditions — Cholangiocarcinoma

STUDY DESIGN:
Intervention Model Description: The subjects with advanced ICC will be treated by HNF4α srRNA intravenously via a peripheral vein.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HNF4α srRNA treatment (Experimental): The subjects with advanced ICC will be treated by HNF4α srRNA intravenously via a peripheral vein.
  According to Amendment 1, the HNF4α srRNA preparation CD-801 used in the original protocol will expire on December 31, 2024. For participants receiving treatment after this date, the preparation will be switched to CD-GA-102, with the treatment dose converted on a 1:1 basis.
  Interventions: Drug: HNF4α srRNA

INTERVENTIONS:
Drug: HNF4α srRNA — HNF4α srRNA will be administered intravenously for the treatment of ICC. The dosing regimen is planned for a second dose 14 ± 3 days post-initial treatment, followed by subsequent treatments every 28 ± 7 days, with adjustments made based on patient tolerance and therapeutic response.
  According to Amendment 1, patients who have received at least 4 cycles of HNF4α srRNA therapy and have a tumor assessment of SD (stable disease) or PD (progressive disease) per RECIST v1.1 criteria may, after a comprehensive evaluation by the investigator considering the patient's treatment history and the current safety and efficacy data of HNF4α srRNA, continue HNF4α srRNA at the same dose, or have their dose adjusted, in combination with immunotherapy, targeted therapy, or chemotherapy.

SUMMARY:
The goal of this investigator-initiated, a single-arm, open-label, pilot study is to investigate the safety, tolerability, and efficacy of intravenous HNF4α srRNA treatment in subjects with advanced Intrahepatic Cholangiocarcinoma (ICC).

Condition of disease: advanced intrahepatic cholangiocarcinoma Intervention： HNF4α srRNA will be administered intravenously for the treatment of ICC. The dosing regimen is planned for a second dose 14 ± 3 days post-initial treatment, followed by subsequent treatments every 28 ± 7 days, with adjustments made based on patient tolerance and therapeutic response. This is a dose escalation assay employing a i3+3 design to assess escalating HNF4α srRNA dosages: 25 μg, 50 μg, and 100 μg. Post-initial dose, a 14-day dose-limiting toxicities (DLT) observation will evaluate tolerability and safety, guiding dose adjustments or selection of the Recommended Dose (RD) for the expansion phase. Cohorts may include up to 9 participants, adjusted for safety.

Drug: HNF4α srRNA, a drug specifically designed to target liver cancer cells and facilitate the expression of HNF4α.

According to Amendment 1, patients who have received at least 4 cycles of HNF4α srRNA therapy and have a tumor assessment of SD (stable disease) or PD (progressive disease) per RECIST v1.1 criteria may, after a comprehensive evaluation by the investigator considering the patient's treatment history and the current safety and efficacy data of HNF4α srRNA, continue HNF4α srRNA at the same dose, or have their dose adjusted, in combination with immunotherapy, targeted therapy, or chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, aged 18 years or older.
2. Histologically or cytologically confirmed intrahepatic cholangiocarcinoma patients.
3. Patients with intrahepatic cholangiocarcinoma not suitable for surgical resection, liver transplantation, or ablation therapy, or those with post-surgical recurrence and/or metastasis.
4. Patients not suitable for local or systemic treatment, or those who have progressed after at least one chemotherapy regimen containing gemcitabine/fluoropyrimidine/platinum, etc..
5. Life expectancy of 12 weeks or more.
6. Subjects must have an Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0 to 2.
7. Males with fertility and females of childbearing potential are willing to use a highly effective method of contraception for the entire study period and for 6 months after study drug discontinuation. Females of childbearing age, including premenopausal females and within 2 years after menopause, must have a negative serum pregnancy test result within 7 days prior to the first dose of study treatment.
8. Subjects who had a voluntary agreement to provide written informed consent and the willingness and ability to comply with all aspects of the protocol.

Exclusion Criteria:

* Patients with any of the following criteria were excluded from participation in this study

  1. Inadequate liver function：Albumin (ALB) < 25 g/L, or total bilirubin > 5 × the upper limit of normal (ULN), or aspartate aminotransferase (AST), alkaline phosphatase (ALP), or alanine aminotransferase (ALT) >10 × ULN.
  2. Inadequate renal function defined as creatinine >1.5 × ULN or calculated creatinine clearance < 40 mL/min.
  3. Absolute neutrophil count (ANC) < 1.0×109/L, or Platelets < 30×109/L, or Hemoglobin < 8.5 g/dL.
  4. International normalized ratio (INR) > 2.3.
  5. Poorly controlled hypertension, diabetes or other serious heart or lung diseases, or with serious dysfunction.
  6. Patients who have received local or systemic anti-tumor treatments such as ablation, Transhepatic Arterial Chemotherapy and Embolization (TACE), local radiotherapy of the liver, immunotherapy, targeted therapy, etc., within 4 weeks, or chemotherapy, other trial drugs, or radiotherapy of metastatic lesions within 2 weeks, except for treatment regimens assessed as disease progression according to RECIST v1.1.
  7. Patients with incurable brain metastasis.
  8. All toxicities related to prior locoregional or systemic anti-tumor treatments are still grade 2 or more (except for hair loss and other events that have been judged tolerable by researchers).
  9. Complication histories of liver cirrhosis or HCC such as gastrointestinal hemorrhage, overt hepatic encephalopathy, or refractory ascites within 2 weeks prior to the first dose of study treatment.
  10. Uncontrolled active infection (eg, lung infections, or abdominal infections).
  11. History of malignancy other than HCC within 5 years prior to screening, with the exception of malignancies with a negligible risk of metastasis or death (e.g., 5-year overall survival rate > 90%), such as adequately treated early gastric carcinoma, carcinoma in situ of the cervix, non-melanoma skin carcinoma, or localized prostate cancer.
  12. Hepatitis B virus DNA greater than 500 copies/mL, or hepatitis C virus RNA greater than 15 U/mL.
  13. Positive for human immunodeficiency virus (HIV).
  14. Allergic to contrast agents.
  15. Pregnant/lactating women, or women with the possibility of pregnancy.
  16. Any medical conditions which, in the opinion of the investigator, would preclude participation in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2024-11-07 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
To evaluate the tolerability and safety for intravenous HNF4α srRNA in subjects with intrahepatic cholangiocarcinoma (ICC) | Through study completion, an average of 2 years
  Safety and tolerability are assessed based on the incidence of Dose-Limiting Toxicities (DLTs) within 14 days post-initial drug administration, along with the frequency and severity of adverse events (AEs), serious adverse events (SAEs), and events leading to treatment discontinuation throughout the treatment period, all evaluated using the Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0. According to Amendment 1, the primary endpoint has been amended from assessing the incidence and severity of DLTs, adverse events (AEs), serious adverse events (SAEs), and AEs leading to treatment discontinuation (evaluated per NCI-CTCAE 5.0) with HNF4α srRNA therapy to assessing these outcomes for both HNF4α srRNA monotherapy and combination therapy.

SECONDARY OUTCOMES:
To assess the objective response rate (ORR) by RECIST v1.1 | From the first study dose date until the date of documented complete response or partial response, assessed up to 24 months.
  To assess the proportion of subjects who have best overall response of complete response or partial response at the time of data cutoff based on RECIST v1.1. According to Amendment 1, the secondary endpoint has been updated from evaluating the ORR per RECIST v1.1 with HNF4α srRNA therapy to evaluating the ORR for both monotherapy and combination therapy with HNF4α srRNA per RECIST v1.1.
Duration of response based on RECIST v1.1 | up to 24 months
  To assess the time from the first documentation of complete response or partial response to the date of first documentation of disease progression or death (whichever occurs first) based on RECIST v1.1
Progression-free survival based on RECIST v1.1 | up to 24 months
  To assess the time from the first study dose date to the date of first documentation of disease progression or death(whichever occurs first) based on RECIST v1.1
Time to response based on RECIST v1.1 | up to 24 months
  To assess the time from the date of first study dose to the date of first documentation of complete response or partial response based on RECIST v1.1
Clinical benefit rate based on RECIST v1.1 | up to 24 months
  To assess the proportion of subjects who have best overall response of complete response or partial response or durable stable disease (duration of stable disease ≥ 23 weeks) based on RECIST v1.1
Overall Survival | Throughout the entire course of treatment until the end of the follow-up period, an average of 2 years
  To assess the time from the first study dose date until date of death from any cause . Subjects who are lost to follow-up and the subjects who are alive at the date of data cutoff will be censored at the date the subject was last known alive or the cut-off date, whichever comes earlier.
Patient Reported Outcome-1 | Through study completion, an average of 2 years
  The effect of HNF4α srRNA on the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30，EORTC QLQ-C30
Patient Reported Outcome-2 | Through study completion, an average of 2 years
  The effect of HNF4α srRNA on the European Organization for Research and Treatment of Cancer Quality of Life, EORTC QLQ-BIL21 Questionnaire-BIL21
Patient Reported Outcome-3 | Through study completion, an average of 2 years
  The effect of HNF4α srRNA on The Generic Euroquol Five Dimension Five Level (EQ-5D-5L) Questionnaire
The impact of HNF4α srRNA treatment on tumor biomarkers in serum | Through study completion, an average of 2 years
  The changes in tumor markers after treatment, including CA19-9, carcinoembryonic antigen (CEA), and alpha-fetoprotein (AFP)

OTHER OUTCOMES:
The assessment of whether the efficacy of HNF4α srRNA is related to specific mutations | Through study completion, an average of 2 years
  Identification of whether the efficacy of HNF4α srRNA is related to specific gene mutations in ICC tissue through next-generation sequencing
The impact of HNF4α srRNA treatment on proteomics in serum | Through study completion, an average of 2 years
  The detection of proteomics in patient serum before and after treatment of HNF4α srRNA
The impact of HNF4α srRNA treatment on metabolomics in serum | Through study completion, an average of 2 years
  The detection of metabolomics in patient serum before and after treatment of HNF4α srRNA
The impact of HNF4α srRNA treatment on cytokines in serum | Through study completion, an average of 2 years
  The detection of cytokines in patient serum before and after treatment of HNF4α srRNA
The impact of HNF4α srRNA treatment on immune cell subsets in serum or tissuses | Through study completion, an average of 2 years
  The detection of immune cell subsets in patient serum or ICC tissues before and after treatment of HNF4α srRNA
The impact of HNF4α srRNA treatment on the quantitative enhancement volume standards of intrahepatic cholangiocarcinoma | Through study completion, an average of 2 years
  The changes in tumor enhancement volume pre- and post-treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Changzheng Hospital, Naval Medical University, Shanghai, Shanghai Municipality, China